CLINICAL TRIAL: NCT06111781
Title: The SUGAR Study: (SBRT and Ultrashort GnRH Antagonist-Relugolix) for Clinicogenomic Unfavorable Intermediate Risk Prostate Cancer
Brief Title: The SUGAR Study; SBRT and Relugolix) for Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000036163; No NIH funding (Other: 10.20.23)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix

STUDY DESIGN:
Intervention Model Description: Participants will undergo baseline tests at the beginning of the study and will be randomized to receive Stereotactic body radiotherapy (SBRT) + Ultrashort GNRH Antagonist Relugolix (SUGAR) vs. Stereotactic body radiotherapy (SBRT) alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stereotactic body radiotherapy (Active Comparator): SBRT Though a range of doses are delivered nationally for IR prostate cancer, the most common regimen is 7.25 Gy- 8.00 Gy x 5 fractions, given over 2 weeks.
  Interventions: Radiation: SBRT standard of care radiotherapy treatment
- Relugolix and SBRT (Active Comparator): SBRT and Relugolix SBRT along with 30 days of total relugolix (study drug) will be used. Relugolix starting 14 days to 17 days prior to the first treatment.
  Interventions: Drug: Relugolix 120 MG [Orgovyx]; Radiation: SBRT standard of care radiotherapy treatment

INTERVENTIONS:
Drug: Relugolix 120 MG [Orgovyx] — ORGOVYX will be initiated with a loading dose of 360 mg on the first day and continue treatment with a 120 mg dose taken orally once daily at approximately the same time each day. Total length of treatment will be 30 days.
  Other Names: SBRT standard of care radiotherapy treatment and Relugolix
  Arms: Relugolix and SBRT
Radiation: SBRT standard of care radiotherapy treatment — SBRT is a standard-of-care radiotherapy treatment for intermediate-risk prostate cancer.

SUMMARY:
The goal of this clinical trial is to measure the toxicity and effectiveness of the following treatments for cFIR/cgUIR prostate cancer patients.

Stereotactic body radiotherapy (SBRT) alone or Stereotactic body radiotherapy (SBRT) combined with Ultrashort GNRH Antagonist called Relugolix (an oral drug). Treatments will be randomly assigned to study patients.

The main questions it aims to answer are the following:

1. Whether the proportion of men who undergo SUGAR have a superior rate of attaining PSA nadir of <= 0.2 compared to SBRT alone, and
2. Whether SUGAR is superior to historical rates of minimal clinically important decline (MCID) in sexual and hormonal function at 6 months for patients undergoing 6 months of androgen deprivation therapy (ADT)

Men aged 18+ with cFIR/cgUIR will be enrolled. Specifically, patients must meet one of the following 2 criteria: 1) Gleason score must be Gleason 3+4 with a PSA < 20 ng/mL, or 2) Gleason 6 (3+3) and PSA > 10 ng/mL and < 20 ng mL.

DETAILED DESCRIPTION:
Unfavorable Intermediate Risk (UIR) Prostate Cancer is prostate cancer that is localized and curable but may require more treatment than external beam radiotherapy (EBRT) alone. In contrast, favorable intermediate risk (FIR) prostate cancer can be treated by EBRT alone. There is evidence that some prostate cancer that is classified through clinical factors as FIR can act more aggressively if also associated with a high risk gene expression score. This type of prostate cancer (traditionally favorable intermediate risk, but with a gene signature that predicts for aggressive disease) presents a treatment dilemma.

Recent evidence suggests that androgen deprivation therapy (ADT) is generally beneficial for intermediate risk prostate cancer and so it is possible that these patients (with favorable intermediate risk based on non-genetic factors but with high genetic risk) may also benefit. However, ADT causes very bothersome side effects including hot flashes, fatigue, sexual disfunction, and in some cases, heart problems. In order to balance the benefit and harms of ADT in combination with radiation, we could reduce the length of ADT and make it precisely overlap with radiation treatment. The oral ADT medication Relugolix (Orgovyx) is ideal for this purpose. In addition to shortening ADT, it is important to measure any potential benefit when ADT is added to stereotactic body radiotherapy (SBRT). SBRT is a shorter and more intense version of standard fractionation EBRT.

Therefore, a multicenter randomized phase III study comparing prostate cancer control and quality of life with SBRT + Ultrashort GNRH Antagonist Relugolix (SUGAR) vs. SBRT alone for a category of clinicogenomic unfavorable intermediate risk patients with favorable clinical features and high risk genetic features.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Has histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
4. Born assigned to Male gender, age 18 and above. Female identifying transgender or gender fluid are allowed on study provided they have not undergone testosterone suppressing therapy and were born with a prostate.
5. Has a serum testosterone at the Screening visit of >150 ng/dL
6. Has a serum PSA concentration at the Screening visit of > 0.2 ng/mL
7. Able to swallow pills and take medication orally (no documented inability to eat solids and swallow pills) and be willing to adhere to the tice daily regimen of medication (if assigned to the experimental arm).
8. For patients of reproductive potential: use of condoms or other methods (including abstinence) to ensure effective contraception with partner during radiotherapy and through 4 months after the last dose of the study drug or radiotherapy
9. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration
10. Clinical favorable intermediate risk prostate cancer: Gleason score must be Gleason 3+4 with a PSA < 20 ng/mL, or Gleason 6 (3+3) and PSA > 10 ng/mL and < 20 ng mL.
11. Decipher GC score of 0.6 or higher or higher indicating high genomic risk for most recent biopsy
12. Documented prostate volume (by MRI or ultrasound) <= 80 cc

Exclusion Criteria:

1. Current use of medications that cause QT prolongation
2. Known allergic reactions to relugolix
3. Treatment with another investigational drug or other intervention for prostate cancer within 30 days of enrollment
4. Ulcerative colitis or other inflammatory bowel disease history
5. Connective tissue disease such as lupus, scleroderma, or dermatomyositis
6. GNRH antagonist therapy or SBRT to the prostate are medically contraindicated or not tolerated
7. History of long QT syndrome documented in the medical record
8. The following ECG abnormalities are excluded:

   1. Q-wave infarction unless identified 6 or more months before the Screening Visit
   2. QT interval corrected for heart rate (QTc) > 470 msec. If the QTc is prolonged in a patient with a pacemaker, the patient may be enrolled in the study upon discussion with the study PI
   3. Congenital long QT syndromeQ
9. History of surgical castration
10. Prior treatment for prostate cancer with surgery or prostate directed radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Born assigned to Male gender
Enrollment: 60 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants that attain PSA nadir | up to 2 years post treatment
  The proportion of men who undergo SUGAR that attain PSA nadir of <= 0.2ng/mL compared to SBRT alone.

SECONDARY OUTCOMES:
Change in Quality of life assessment using the EPIC-26 survey | up to 2 years post treatment
  The EPIC-26 is a validated instrument that measures health-related quality of life over 5 domains: Urinary incontinence, Urinary irritative/obstructive, Bowel, Sexual, Hormonal. Range of scores are 0-100. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: James Yu, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No